CLINICAL TRIAL: NCT02658825
Title: A Double-blind, Double-dummy, Randomized, 3-Period Cross-over, Placebo- and Positive-controlled Study to Evaluate the Effect of JNJ-63623872 on Cardiac Repolarization Interval in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of JNJ-63623872 on Cardiac Repolarization Interval in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR108108; 63623872FLZ1005 (Other: Janssen Research & Development, LLC); 2015-004365-82 (EudraCT Number)
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy; JNJ-63623872; Moxifloxacin
MeSH Terms: interventions — pimodivir; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Panel 1: Dose level 1 (Experimental): Participants will receive either treatment A (JNJ-63623872, 2400 milligram (mg) tablet orally once on Day 1) or treatment B [(placebo (matching with JNJ-63623872 2400 mg) tablet orally once on Day 1].
  Interventions: Drug: JNJ-63623872 2400 milligram (mg); Drug: Placebo (Matching with JNJ-63623872 2400 mg)
- Panel 1: Dose level 2 (Experimental): Participants will receive either treatment C (JNJ-63623872, 3000 mg tablet orally once on Day 1) or treatment D [placebo (matching with JNJ-63623872 3000 mg) tablet orally once on Day 1].
  Interventions: Drug: JNJ-63623872 3000 mg; Drug: Placebo (Matching with JNJ-63623872 3000 mg)
- Panel 2: Treatment EFG (Experimental): Participants will receive treatment E (JNJ-63623872 dose selected in Panel 1 tablet and placebo matching with moxifloxacin) in Period 1; followed by treatment F (placebo matching with JNJ-63623872 and moxifloxacin 400 mg capsule) in Period 2; followed by treatment G (placebo matching with JNJ-63623872 and placebo matching with moxifloxacin) in Period 3. A washout period of 5 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-63623872; Drug: Moxifloxacin; Drug: Placebo (Matching with JNJ-63623872 Dose); Drug: Placebo (Matching with Moxifloxacin)
- Panel 2: Treatment FGE (Experimental): Participants will receive treatment F (placebo matching with JNJ-63623872 and moxifloxacin 400 mg capsule) in Period 1; followed by treatment G (placebo matching with JNJ-63623872 and placebo matching with moxifloxacin) in Period 2; followed by treatment E (JNJ-63623872 dose selected in Panel 1 tablet and placebo matching with moxifloxacin) in Period 3. A washout period of 5 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-63623872; Drug: Moxifloxacin; Drug: Placebo (Matching with JNJ-63623872 Dose); Drug: Placebo (Matching with Moxifloxacin)
- Panel 2: Treatment GEF (Experimental): Participants will receive treatment G (placebo matching with JNJ-63623872 and placebo matching with moxifloxacin) in Period 1; followed by treatment E (JNJ-63623872 dose selected in Panel 1 tablet and placebo matching with moxifloxacin) in Period 2; followed by treatment F (placebo matching with JNJ-63623872 and moxifloxacin 400 mg capsule) in Period 3. A washout period of 5 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-63623872; Drug: Moxifloxacin; Drug: Placebo (Matching with JNJ-63623872 Dose); Drug: Placebo (Matching with Moxifloxacin)
- Panel 2: Treatment GFE (Experimental): Participants will receive treatment G (placebo matching with JNJ-63623872 and placebo matching with moxifloxacin) in Period 1; followed by treatment F (placebo matching with JNJ-63623872 and moxifloxacin 400 mg capsule) in Period 2; followed by treatment E (JNJ-63623872 dose selected in Panel 1 tablet and placebo matching with moxifloxacin) in Period 3. A washout period of 5 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-63623872; Drug: Moxifloxacin; Drug: Placebo (Matching with JNJ-63623872 Dose); Drug: Placebo (Matching with Moxifloxacin)
- Panel 2: Treatment FEG (Experimental): Participants will receive treatment F (placebo matching with JNJ-63623872 and moxifloxacin 400 mg capsule) in Period 1; followed by treatment E (JNJ-63623872 dose selected in Panel 1 tablet and placebo matching with moxifloxacin) in Period 2; followed by treatment G (placebo matching with JNJ-63623872 and placebo matching with moxifloxacin) in Period 3. A washout period of 5 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-63623872; Drug: Moxifloxacin; Drug: Placebo (Matching with JNJ-63623872 Dose); Drug: Placebo (Matching with Moxifloxacin)
- Panel 2: Treatment EGF (Experimental): Participants will receive treatment E (JNJ-63623872 dose selected in Panel 1 tablet and placebo matching with moxifloxacin) in Period 1; followed by treatment G (placebo matching with JNJ-63623872 and placebo matching with moxifloxacin) in Period 2; followed by treatment F (placebo matching with JNJ-63623872 and moxifloxacin 400 mg capsule) in Period 3. A washout period of 5 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-63623872; Drug: Moxifloxacin; Drug: Placebo (Matching with JNJ-63623872 Dose); Drug: Placebo (Matching with Moxifloxacin)

INTERVENTIONS:
Drug: JNJ-63623872 2400 milligram (mg) — Participants will receive JNJ-63623872 2400 mg tablet orally once on Day 1 of Panel 1.
  Arms: Panel 1: Dose level 1
Drug: JNJ-63623872 3000 mg — Participants will receive JNJ-63623872 3000 mg tablet orally once on Day 1 of Panel 1.
  Arms: Panel 1: Dose level 2
Drug: JNJ-63623872 — Participants will receive JNJ-63623872 dose selected in Panel 1 tablet orally once on Day 1 of Panel 2.
  Arms: Panel 2: Treatment EFG; Panel 2: Treatment EGF; Panel 2: Treatment FEG; Panel 2: Treatment FGE; Panel 2: Treatment GEF; Panel 2: Treatment GFE
Drug: Moxifloxacin — Participants will receive moxifloxacin 400 mg capsule orally once on Day 1 of Panel 2.
  Arms: Panel 2: Treatment EFG; Panel 2: Treatment EGF; Panel 2: Treatment FEG; Panel 2: Treatment FGE; Panel 2: Treatment GEF; Panel 2: Treatment GFE
Drug: Placebo (Matching with JNJ-63623872 2400 mg) — Participants will receive placebo (matching with JNJ-63623872 2400 mg) tablet orally once on Day 1 of Panel 1.
  Arms: Panel 1: Dose level 1
Drug: Placebo (Matching with JNJ-63623872 3000 mg) — Participants will receive placebo (matching with JNJ-63623872 3000 mg) tablet orally once on Day 1 of Panel 1 and 2.
  Arms: Panel 1: Dose level 2
Drug: Placebo (Matching with JNJ-63623872 Dose) — Participants will receive placebo (matching with JNJ-63623872 dose) tablet orally once on Day 1 of Panel 2.
  Arms: Panel 2: Treatment EFG; Panel 2: Treatment EGF; Panel 2: Treatment FEG; Panel 2: Treatment FGE; Panel 2: Treatment GEF; Panel 2: Treatment GFE
Drug: Placebo (Matching with Moxifloxacin) — Participants will receive placebo (matching with Moxifloxacin) tablet orally once on Day 1 of Panel 2.
  Arms: Panel 2: Treatment EFG; Panel 2: Treatment EGF; Panel 2: Treatment FEG; Panel 2: Treatment FGE; Panel 2: Treatment GEF; Panel 2: Treatment GFE

SUMMARY:
The purpose of this study is to evaluate the effect of JNJ-63623872 on the QT/QTc interval at supratherapeutic exposure in healthy participants (Panel 2).

DETAILED DESCRIPTION:
This is a two-part Phase 1 study consisting of a dose escalation part (Panel 1) and a thorough QT (TQT) part (Panel 2). Panel 1 will be a double-blind (neither the researchers nor the participants know what treatment the participant is receiving), randomized (study medication assigned to participants by chance), placebo-controlled dose escalation study in healthy participants to determine the safety, tolerability and pharmacokinetics of JNJ-63623872 after administration of single doses of 2400 milligrams (mg) and 3000 mg under fasted conditions. The final dose to be used in the Panel 2 will be determined based on the results of this dose escalation part. An interim analysis will be conducted on Panel 1 to select the dose for Panel 2. Panel 2 will be a double-blind, double-dummy, randomized, 3-period crossover (the same medications provided to all participants but in different sequence), placebo- and positive controlled study to evaluate the effect of JNJ-63623872 on the QT/QTc interval in healthy participants. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Each participant must sign an Informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and is willing to participate in the study
* Participant must be willing and able to adhere to the prohibitions and restrictions specified in the protocol
* A female participant must agree not to donate eggs (ova, oocytes) during the study and for at least 90 days after receiving the (last dose of) study drug
* A male participant who is sexually active with a woman of childbearing potential must agree to use two effective methods of contraception during the study and for at least 90 days after receiving the (last dose of) study drug, and a male participant must also not donate sperm during the study and for at least 90 days after receiving the (last dose of) study drug
* Participants must be non-smokers for at least 3 months prior to Screening
* Participants must have a Body Mass Index (BMI) between 18.0 and 30.0 kilogram per meter^2 (kg/m^2) (inclusive) at Screening

Exclusion Criteria:

* Participant has a history of current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the Investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Participants with a history of clinically relevant heart rhythm disturbances including atrial, junctional, re-entry, and ventricular tachycardias, and heart blocks
* Participants with unusual T wave morphology (such as bifid T wave) likely to interfere with QTc measurements
* Participants with electrolyte abnormalities (hypokalemia, hypocalcemia, hypomagnesemia) of grade 2 or above within 21 days prior to the (first) intake of the study drug
* Participants with a breast implant or a history of thoracic surgery likely to cause abnormality of the electrical conduction through thoracic tissues
* Participant has taken any disallowed therapies (Concomitant Therapy) before the planned (first) intake of study drug
* Participant has known allergies, hypersensitivity, or intolerance to JNJ-63623872, moxifloxacin or its excipients

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2016-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Corrected QT Interval (QTc) at Different Time Points | 45, 30 and 15 minutes predose and 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hours postdose on Day 1
  Electrocardiogram will be collected by Holter monitoring. The measured QT data will be corrected for heart rate using Fridericia (QTcF), Bazett (QTcB), and study-specific power (QTcP) correction methods. The QTcF as primary correction method.

SECONDARY OUTCOMES:
Maximum Observed Concentration (Cmax) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 120 hours post-dose on Day 1 of Treatment A of Dose Level 1, Treatment C of Dose Level 2 (Panel 1) and Treatment E (Panel 2)
  The Cmax is the maximum observed concentration.
Time To Reach The Maximum Observed Concentration (Tmax) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 120 hours post-dose on Day 1 of Treatment A of Dose Level 1, Treatment C of Dose Level 2 (Panel 1) and Treatment E (Panel 2)
  The Tmax is the actual sampling time to reach the maximum observed concentration.
Observed Concentration at 24 Hours Post Dosing (C24h) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 120 hours post-dose on Day 1 of Treatment A of Dose Level 1, and Treatment C of Dose Level 2 (Panel 1)
  The C24h is the observed concentration at 24 hours post dosing.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 120 hours post-dose on Day 1 of Treatment A of Dose Level 1, and Treatment C of Dose Level 2 (Panel 1)
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time 0 to Infinite Time (AUC[0-infinity]) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 120 hours post-dose on Day 1 of Treatment A of Dose Level 1, and Treatment C of Dose Level 2 (Panel 1)
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Area Under the Concentration Versus Time Curve (AUC) From Time of Administration up to 24 Hours Post Dosing (AUC24h) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose on Day 1 of Treatment E (Panel 2)
  The AUC24h is the area under the concentration versus time curve (AUC) from time of administration up to 24 hours post dosing.
Elimination Rate Constant (Lambda[z]) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 120 hours post-dose on Day 1 of Treatment A of Dose Level 1, and Treatment C of Dose Level 2 (Panel 1)
  Lambda (z) is first-order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Apparent Terminal Elimination Half-life (t1/2term) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 120 hours post-dose on Day 1 of Treatment A of Dose Level 1, and Treatment C of Dose Level 2 (Panel 1)
  The T1/2term is the apparent terminal elimination half-life, calculated as 0.693/Lambda(z).
Number of Participants with Adverse Events (AEs) and Serious AEs | Screening up to Follow-up (10 to 14 days after last study drug administration)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Antwerp, Belgium